CLINICAL TRIAL: NCT04908826
Title: Comparison of Administration of Indocyanine Green (ICG) for Image-Guided Laparoscopic Cholocystectomy- A Randomized, Controlled, Prospective Trial
Brief Title: Comparison of Icg's Route of Administration During Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Savvas Simeonidis, Principal Investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3765/03.02.2020
Record Dates: First submitted 2021-05-10; First posted 2021-06-01 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Laparoscopic; Cholecystectomy; Cholelithiasis; Bile Duct; Choledocholithiasis; Stone - Biliary; Post-Op Complication; Cholangiography; Indocyanine Green; Intraoperative Complications; Bile Duct Injury
MeSH Terms: conditions — Cholelithiasis; Choledocholithiasis; Cholecystolithiasis; Postoperative Complications; Intraoperative Complications | interventions — Indocyanine Green; Organization and Administration; Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (standard cholangiography during surgery) (Active Comparator): All patients will undergo laparoscopic cholecystectomy. In this group standard cholangiography will be performed during surgery. Standard cholangiography will be performed with selective catheterization of the cystic duct and infusion of a radiolucent substance (non-ionic low osmotic iodine). The category includes drugs such as iohexol, iopamidol, iopromide, ioversol, iobitriol, iomeprol and iodixanol. In our study we will use Xenetix (iobitriol) and perform cholangiography with C-ARM recording.
  Interventions: Procedure: Indocyanine Green (ICG) administration
- Group B (cholangiography with iv administration of icg prior to surgery) (Active Comparator): All patients will undergo laparoscopic cholecystectomy. In this group intravenous fluorescent cholangiography with indocyanine green will be given at a dose of 0.3 mg / mL / Kg 6 (six) hours before the start of surgery.The bile duct system will be recorded with a special camera (Karl Storz NIR / ICG).
  Interventions: Procedure: Indocyanine Green (ICG) administration
- Group C (cholangiography with direct administration of icg to the bile duct system during surgery) (Active Comparator): All patients will undergo laparoscopic cholecystectomy. In the third group intraoperative cholangiography will be performed with direct administration of indocyanine green at a dose of 0.03 mg / ml / Kg to the bile duct cyst.
  Interventions: Procedure: Indocyanine Green (ICG) administration

INTERVENTIONS:
Procedure: Indocyanine Green (ICG) administration — Patients will undergo laparoscopic cholecystectomy after they are randomly divided into 3 (three) groups. A total of 240 patients will be randomized into three groups of 80. In the first group (A) standard cholangiography will be performed. In group (B) intravenous fluorescent cholangiography with indocyanine green will be performed during surgery. ICG at a dose of 0.3 mg / mL / Kg 6 (six) hours prior to surgery will be administered. In the third group (C), intraoperative cholangiography will be performed with direct administration of indocyanine green at a dose of 0.03 mg / ml / Kg to the gallbladder.
  Other Names: laparoscopic cholecystectomy; intra-operative cholangiography; c-arm recording; iodine solution administration

SUMMARY:
The aim of the trial is to compare the routes of administration of indocyanine green (ICG) during laparoscopic cholocystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is now the method of choice for the treatment of symptomatic and complicated gallstones.

There are two major problems that can occur during and after a laparoscopic cholecystectomy. These are the remaining stones in the bile duct and the iatrogenic injuries of the bile ducts. Iatrogenic bile duct injuries are the most difficult complication of cholecystectomy and are a clinical entity that needs multifactorial treatment as it significantly increases morbidity, mortality and overall cost. Intraoperative cholangiography is used to prevent these complications.

Intraoperative cholangiography is the traditional method of identifying bile duct anatomy during laparoscopic cholecystectomy. This method has the disadvantages that both the patient and the staff are exposed to radiation, while in order to perform it, catheterization of the cystic duct must be performed, which requires surgical procedures that increase the time of the operation, while in some cases it is not technically easy. Finally, with the intraoperative cholangiography, the injuries of the bile ducts are detected, after they have taken place, therefore it helps in their timely diagnosis but does not limit the frequency of their occurrence.

Indocyanine green is a sterile, anionic, water-soluble but relatively hydrophobic tricarbocyanine molecule with a molecular weight of 751.4. It was developed in 1955 at Kodak Laboratories and in 1959 was approved for clinical use by the FDA. It has the property of fluorescing, after its administration, with a maximum absorption at 800 nm after exposure to infrared lighting. Its use offers an image of high clarity and sensitivity, target imaging, with parallel low acoustic emission. Indocyanine green has the following properties and advantages, which make it an important tool in the applications of medical sciences and studies.

Following intravenous administration, it binds to plasma lipoproteins with minimal escape into the interstitial space. Extremely important for its clinical use is the complete excretion through the bile, as well as the non-production of metabolic products. It has low toxicity in the absence of ionization, which in combination with the short half-life of the substance, provides safety for the patient in its use and application in medical and biomedical sciences. It has low costs that in combination with its ease of use facilitates its application. No expensive equipment or large learning curve required. Also the possibility of recurrence with re-administration intraoperatively can offer a number of applications in laparoscopic surgery. It has a low rate of side effects and interactions with other drugs and preparations, a major allergic reaction has been reported in the literature. The first clinical applications of indocyanine green were to assess cardiac function, liver function in cirrhotic patients before hepatectomy, and to examine the retinal vessels.

Its use in laparoscopic cholecystectomy, as already mentioned, is based on its ability to fluoresce when exposed to infrared light and in combination with the fact that when administered intravenously it is concentrated and excreted from the bile offers the possibility of intraoperative, fluorescent cholangiography that aims to identify the elements of the Callot triangle.

This study aims to demonstrate that endocyanin green cholangiography is equivalent to or better than conventional cholangiography for the diagnosis of cholelithiasis and biliary injuries. It is therefore an important clinical application that will probably facilitate surgeons both in the prevention of biliary injuries and in the intraoperative diagnosis of cholelithiasis.

Patients who will undergo laparoscopic cholecystectomy will be randomly divided into 3 (three) groups. The processing of the results will be done in the appropriate way and method. A total of 240 patients will be randomized into three groups of 80. In the first group (A) classical cholangiography will be performed. In group (B) will be performed intravenous fluorescent cholangiography with indocyanine green 6 (six) hours before the start of surgery. In the third group (C) will be performed intraoperative cholangiography with direct administration of indocyanine green to the gallbladder.

ELIGIBILITY:
Inclusion Criteria:

1. age older than 18 years old
2. laparoscopic cholecystectomy
3. elective surgery

Exclusion Criteria:

1. younger than 18 years old
2. no consent to participate to the study
3. history of allergic reaction to iodine products
4. urgent or emergent cholecystectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
successful imaging of biliary system | intra-operatively
  The anatomy of the extrahepatic bile ducts will be orally determined by the surgeon and the cases in which the oral description will coincide with the findings of cholangiography or not and where there were differences will be recorded.
operation duration | intra-operatively
  minutes
intra-operative complications (bleeding, bile duct leakage, bile duct injury) | intra-operatively
  presence or absence
applicability of the intra-operatively cholangiography | intra-operatively
  yes or no
presence of bile duct stones (choledocholithiasis) | intra-operatively
  yes or no

SECONDARY OUTCOMES:
gender | pre-operatively
  male or female
ASA score | pre-operatively
  number
age | pre-operatively
  years
body mass index | pre-operatively
  kg/m2
indication for laparoscopic cholecystectomy | pre-operatively
  yes or no
SGOT | 24 hours prior to surgery and 24 hours after the surgery
  g/dL
SGPT | 24 hours prior to surgery and 24 hours after the surgery
  g/dL
ALP | 24 hours prior to surgery and 24 hours after the surgery
  g/dL
γ-GT | 24 hours prior to surgery and 24 hours after the surgery
  g/dL
total bilirubin | 24 hours prior to surgery and 24 hours after the surgery
  mg/dL
indirect bilirubin | 24 hours prior to surgery and 24 hours after the surgery
  mg/dL
direct bilirubin | 24 hours prior to surgery and 24 hours after the surgery
  mg/dL
PT | 24 hours prior to surgery and 24 hours after the surgery
  seconds
INR | 24 hours prior to surgery and 24 hours after the surgery
  number
aPTT | 24 hours prior to surgery and 24 hours after the surgery
  seconds
urea | 24 hours prior to surgery and 24 hours after the surgery
  mg/dL
creatinine | 24 hours prior to surgery and 24 hours after the surgery
  mg/dL
CRP | 24 hours prior to surgery and 24 hours after the surgery
  mg/L
WBC | 24 hours prior to surgery and 24 hours after the surgery
  mm3/L
ESR | 24 hours prior to surgery and 24 hours after the surgery
  mm
procalcitonin | 24 hours prior to surgery and 24 hours after the surgery
  mg/dL
TNF-a | 24 hours prior to surgery and 24 hours after the surgery
  pg/ml
IL-6 | 24 hours prior to surgery and 24 hours after the surgery
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Savvas Simeonidis, MD, PhD(c), Principal Investigator — General Hospital of Thessaloniki "G. Papanikolaou", Aristotle University of Thessaloniki
Locations (1):
- General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costi R, Gnocchi A, Di Mario F, Sarli L. Diagnosis and management of choledocholithiasis in the golden age of imaging, endoscopy and laparoscopy. World J Gastroenterol. 2014 Oct 7;20(37):13382-401. doi: 10.3748/wjg.v20.i37.13382. PMID 25309071
- [Background] Duca S, Bala O, Al-Hajjar N, Lancu C, Puia IC, Munteanu D, Graur F. Laparoscopic cholecystectomy: incidents and complications. A retrospective analysis of 9542 consecutive laparoscopic operations. HPB (Oxford). 2003;5(3):152-8. doi: 10.1080/13651820310015293. PMID 18332976
- [Background] Al-Mulhim AA. Current trends in laparoscopic cholecystectomy. J Family Community Med. 1997 Jul;4(2):33-40. PMID 23008571
- [Background] Duncan CB, Riall TS. Evidence-based current surgical practice: calculous gallbladder disease. J Gastrointest Surg. 2012 Nov;16(11):2011-25. doi: 10.1007/s11605-012-2024-1. Epub 2012 Sep 18. PMID 22986769
- [Background] Alander JT, Kaartinen I, Laakso A, Patila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585. doi: 10.1155/2012/940585. Epub 2012 Apr 22. PMID 22577366
- [Background] Boni L, David G, Mangano A, Dionigi G, Rausei S, Spampatti S, Cassinotti E, Fingerhut A. Clinical applications of indocyanine green (ICG) enhanced fluorescence in laparoscopic surgery. Surg Endosc. 2015 Jul;29(7):2046-55. doi: 10.1007/s00464-014-3895-x. Epub 2014 Oct 11. PMID 25303914
- [Background] Ambe PC, Plambeck J, Fernandez-Jesberg V, Zarras K. The role of indocyanine green fluoroscopy for intraoperative bile duct visualization during laparoscopic cholecystectomy: an observational cohort study in 70 patients. Patient Saf Surg. 2019 Jan 12;13:2. doi: 10.1186/s13037-019-0182-8. eCollection 2019. PMID 30651756
- [Background] Chu W, Chennamsetty A, Toroussian R, Lau C. Anaphylactic Shock After Intravenous Administration of Indocyanine Green During Robotic Partial Nephrectomy. Urol Case Rep. 2017 Mar 10;12:37-38. doi: 10.1016/j.eucr.2017.02.006. eCollection 2017 May. PMID 28316935
- [Background] Hope-Ross M, Yannuzzi LA, Gragoudas ES, Guyer DR, Slakter JS, Sorenson JA, Krupsky S, Orlock DA, Puliafito CA. Adverse reactions due to indocyanine green. Ophthalmology. 1994 Mar;101(3):529-33. doi: 10.1016/s0161-6420(94)31303-0. PMID 8127574